CLINICAL TRIAL: NCT01247922
Title: Open-label Phase 2 Study of Single-agent Erlotinib for Patients With Pediatric Ependymoma Previously Treated With Oral Etoposide in Protocol OSI-774-205
Brief Title: Single-agent Erlotinib in Patients Previously Treated With Oral Etoposide in Protocol OSI-774-205
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: In a pre-planned interim analysis, OSI-774-205 met futility for efficacy with no safety concerns. As a result, the companion trial, OSI-774-206 has been stopped
Sponsor: OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSI-774-206; 2010-023478-38 (EudraCT Number)
Record Dates: First submitted 2010-11-23; First posted 2010-11-25 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Ependymoma
Keywords: Pediatric Ependymoma; Ependymoma; Tarceva; Erlotinib
MeSH Terms: conditions — Ependymoma; Familial ependymoma | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Erlotinib (Experimental): Participants who received erlotinib in a continuous oral dose of 85 mg/m^2 per day until dose modification, interruption or study discontinuation occurred.
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — continuous oral Erlotinib 85 mg/m^2 per day
  Other Names: Tarceva; OSI-774

SUMMARY:
Participants that were assigned to the oral etoposide treatment arm in protocol OSI-774-205 and either progressed while on study or discontinued due to unacceptable toxicity related to etoposide were allowed to participate in this study to assess the safety profile of single-agent erlotinib in participants with recurrent or refractory pediatric ependymoma.

DETAILED DESCRIPTION:
The protocol-specified futility criteria were met at the second interim analysis dated 15 Aug 2012 for OSI-774-205. Per the Data Monitoring Committee's recommendation and FDA's agreement, the enrollment of patients in that study and Study OSI-774-206 was permanently closed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been enrolled in OSI-774-205, been randomized to oral etoposide and either progressed while on study or discontinued due to unacceptable toxicity related to etoposide
* Performance status: Lansky ≥ 50% for patients ≤ 10 years of age or younger or Karnofsky ≥ 50% for patients greater than 10 years of age
* Patients must have recovered from any acute toxicity to any prior anti-cancer treatment
* Total bilirubin ≤ 1.5 x upper limit of normal (ULN) for age, serum glutamic pyruvic transaminase (SGPT) ALT ≤ 3 x ULN
* Serum creatinine based on age OR Creatinine Clearance/Glomerular Filtration Rate (GFR) ≥ 70 mL/min/m2
* Patients must be neurologically stable for at least 7 days before registration
* Patients, both males and females, with reproductive potential must agree to practice effective contraceptive measures for the duration of study drug therapy and for at least 90 days after completion of study drug therapy
* Patients must be able to take erlotinib orally

Exclusion Criteria:

* Taking strong/moderate CYP3A4 or CYP1A2 inhibitors/inducers ≤ 14 days before registration
* Have received any other chemotherapy or immunotherapy to treat ependymoma after discontinuation from OSI-774-205
* Taking proton pump inhibitors ≤ 14 days before registration
* Participating in another investigational drug trial while on study
* Pregnant or breast-feeding

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2012-09-13 (Actual); Study Completion 2012-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Astellas Pharma Global Development
Locations (21):
- United States (11):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Children's Hospital of Orange County (CHOC), Orange, California
  - Packard Children's Hospital, Palo Alto, California
  - The Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Children's National Medical Center -D.C. Center for Cancer and Blood Disorders, Washington D.C., District of Columbia
  - University of Miami, Miami, Florida
  - Emory University Children's Healthcare of Atlanta, Atlanta, Georgia
  - University of Minnesota - Amplatz Children's Hospital, Minneapolis, Minnesota
  - Oregon Health & Sciences University Doernbecher Children's Hospital, Portland, Oregon
  - Childrens Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin
- Canada (3):
  - Stollery Children's Hospital, Edmonton, Alberta
  - Children's and Women's Health Center of BC, Vancouver, British Columbia
  - Hospital for Sick Children, Toronto, Ontario
- United Kingdom (7):
  - Birmingham Children's Hospital Oncology Department, Birmingham
  - Royal Hospital for Sick Children, Glasgow
  - Paediatric Oncology and Haematology Offices,, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Royal Manchester Children's Hospital Ward 84, Manchester
  - University of Nottingham, Nottingham
  - Royal Marsden Hospital, Sutton

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited for this OSI-774-206 study were participants with pediatric ependymoma previously treated with oral etoposide in Study OSI-774-205 who progressed while on study or discontinued due to unacceptable toxicity.
Pre-assignment Details: Participants who consented to enter this OSI-774-206 study and fulfilled all the eligibility criteria (no more than 14 days prior to registration) were enrolled in this study no more than 21 days from the last dose of oral etoposide in Study OSI-774-205.
Period: Overall Study
Arm/Group | Erlotinib
Started | 4
Treated | 4
Completed | 0
Not Completed | 4
Not completed — Disease progression | 4

BASELINE CHARACTERISTICS:
Arm/Group | Erlotinib
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 3
  Asian-Indian subcontinent | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety Assessed Through Evaluation of Physical Examinations, Vital Signs, Clinical Laboratory Tests, and Adverse Events (AEs)
Description: Safety is monitored through AEs, which includes abnormal or clinically significant vital sign assessments, laboratory test, physical examination findings associated with signs and/or symptoms requiring withdrawal, dose modification or medical intervention. A treatment-emergent adverse event (TEAE) was defined as an adverse event observed after starting administration of the study drug. An AE was considered serious (SAE) if it resulted in death, a life-threatening situation, inpatient hospitalization or prolongation of an existing hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect in the offspring of a patient who received study drug or other important medical events.
Time Frame: From first dose of study drug to 30 days after last dose of study drug (The mean treatment duration was 170.5 days)
Population: The analysis population is the Safety Analysis Set (SAF) consisted of all enrolled patients who received at least 1 dose of study drug.
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 4
participants
  Any TEAE | 4
  With at least 1 SAE | 2
  With at least 1 treatment-related SAE | 0
  Discontinued study due to treatment-related AEs | 0
  Died on treatment or within 30 days | 1

2. Secondary Outcome: Best Overall Response
Description: Best overall response was derived from an integrated clinical assessment by the study investigator as per institutional standards. This included radiographic assessments deemed appropriate by the investigator in the normal care of the patient. A determination of best overall response at the end of study treatment (complete response, partial response, minor response or stable disease) was only made if (1) any disease-related neurologic symptoms were stable or improving over the interval of the radiographic assessment and (2) corticosteroid dosing for the control of tumor-related signs/symptoms was stable or decreasing.If the investigator deems that a radiographic assessment is not needed, then evidence of clinical improvement may be used to determine best response provided that corticosteroid dosing for tumor-related signs/symptoms is stable or decreasing.
Time Frame: End of treatment (The mean treatment duration was 170.5 days.)
Population: SAF
Measure: Number; unit: participants
Arm/Group | Erlotinib
Number analyzed (Participants) | 4
participants
  Complete response | 0
  Partial response | 0
  Minor response | 0
  Stable disease | 2
  Disease progression | 2

3. Secondary Outcome: Median Treatment Duration
Time Frame: From first dose of study drug up to last dose of study drug (The mean treatment duration was 170.5 days)
Population: SAF
Measure: Median (Full Range); unit: days
Arm/Group | Erlotinib
Number analyzed (Participants) | 4
days | 91.0 [27 to 473]

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 30 days after last dose of study drug (The mean treatment duration was 170.5 days.)
Arm/Group | Erlotinib
Serious Adverse Events (participants affected / at risk) | 2/4
Other Adverse Events (participants affected / at risk) | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=4)
Convulsion (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
VIIth nerve paralysis (Nervous system disorders) | 1
Brain death (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=4)
Peripheral coldness (Vascular disorders) | 1
Blood bilirubin increased (Investigations) | 1
Weight decreased (Investigations) | 1
Weight increased (Investigations) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2
Dysarthria (Nervous system disorders) | 1
Headache (Nervous system disorders) | 3
Partial seizures (Nervous system disorders) | 1
Vision blurred (Eye disorders) | 1
Fatigue (General disorders) | 3
Pain (General disorders) | 1
Pyrexia (General disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin striae (Skin and subcutaneous tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Posture abnormal (Musculoskeletal and connective tissue disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Nasopharyngitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication for review and comment. Sponsor may delay the publication for an additional to 60 days to seek patent protection.